CLINICAL TRIAL: NCT06489301
Title: Mechanisms for Laser-Induced Rejuvenation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wright State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2023-312
Record Dates: First submitted 2024-05-21; First posted 2024-07-05 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Intervention Model Description: All subjects will receive fractionated laser resurfacing.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Fractionated Laser Resurfacing (Experimental): At 14 days prior to scheduled surgery a 5x5cm square on the left abdomen within the region of skin to be excised and treated with fractionated laser resurfacing. Then at 7 days prior to scheduled surgery a 5 cm diameter circle on the right abdomen within the region of skin to be excised, at least 10 cm away from the square, is treated with fractionated laser resurfacing.
  Interventions: Device: Fractionated Laser Resurfacing

INTERVENTIONS:
Device: Fractionated Laser Resurfacing — A rejuvenating laser that makes tiny holes in the very superficial part of the skin.

SUMMARY:
It has shown that laser wounding of geriatric skin protects it against skin cancer. The purpose of this study is to determine the origin of cells called fibroblasts which are present after treatment with Fractionated Laser Resurfacing (FLR). These cells restore a youth-like ultraviolet B (UVB) response, but where they come from is currently unknown. The study recruits subjects who are scheduled to undergo abdominoplasties to investigate the origin of those cells stimulated by laser treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females 18 and older
* Able to comprehend procedures and risks
* Planning to undergo abdominoplasty surgery
* Minimum amount of skin to be removed is 50 x 20cm

Exclusion Criteria:

* Medical history of not well-controlled diabetes. This is defined as a subject who needs high doses of insulin, recent history of hospitalization for diabetes-related complications, or poor wound health as evidenced by diabetic ulcers. Subjects who have been deemed healthy enough for abdominoplasty surgery would tend to suggest that their diabetes should not be an issue. However, if the subjects have diabetic complications as outlined above, they could affect the wound healing which is the object of this protocol so they would be excluded.
* Pregnant or nursing
* History of pathologically abnormal wound healing such as keloidal scars
* Existing tattoos on the abdomen that are so extensive that they could interfere with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
To test if the new fibroblasts that develop in response to fractionated laser resurfacing (FLR) wounding are derived from blood-derived monocytes. | 2 weeks prior to skin removal and 1 week prior to skin removal
  Identify cells in the skin that have been wounded by FLR at 2 weeks and 1 week previously, for cells that co-express markers for both fibroblasts and monocytes by using single cell RNA-sequencing
To test if possible cells transitioning from monocytes to fibroblasts are found in the top part of the dermis (papillary dermis). | 2 weeks prior to skin removal and 1 week prior to skin removal
  Using tissue RNA-seq, PI will define if co-expressing cells are in the papillary dermis.

SECONDARY OUTCOMES:
To define the number and types of cells populating the skin following fractionated laser resurfacing (FLR) wounding | 2 weeks prior to skin removal and 1 week prior to skin removal
  Define the number and types of cells following FLR wounding at 2 weeks and 1 week prior to skin removal by using single-cell RNA-seq.
To define the locations of the number of cells populating in the skin following fractionated laser resurfacing (FLR) wounding | 2 weeks prior to skin removal and 1 week prior to skin removal
  Define the locations of the number cell following FLR wounding at 2 weeks and 1 week prior to skin removal by using tissue RNA-seq.
To define the locations of the types of cells populating in the skin following fractionated laser resurfacing (FLR) wounding | 2 weeks prior to skin removal and 1 week prior to skin removal
  Define the locations of the different cell types following FLR wounding at 2 weeks and 1 week prior to skin removal by using tissue RNA-seq.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Travers, MD, PhD, Principal Investigator — Wright State University
Locations (1):
- Wright State Physicians, Fairborn, Ohio, United States